CLINICAL TRIAL: NCT05363488
Title: A Retrospective Observational Research Study to Describe the Real World Use of Bosutinib in a Single Centre in Scotland
Brief Title: Retrospective Observational Research Study to Describe the Real World Use of Bosutinib in a Single Centre in Scotland
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1871058; BOSISCOT (Other: Alias Study Number)
Record Dates: First submitted 2022-03-15; First posted 2022-05-06 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Myeloid Leukemia
Keywords: Philadelphia chromosome; Breakpoint Cluster Region/ Abelson (BCR/ABL1); retrospective; observational; chromic myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid; Philadelphia Chromosome | interventions — bosutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Chronic Myeloid Leukaemia: Patients diagnosed with chronic myeloid leukaemia treated with Bosutinib
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib — Patients receiving bosutinib treatment
  Other Names: Bosulif

SUMMARY:
This study will describe the efficacy and safety of bosutinib in patients with chronic myeloid leukaemia (CML) used in a real world clinical practice setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Ph+ CML aged ≥18 years at bosutinib initiation.
* Patients prescribed bosutinib (irrespective of the phase of their disease) EITHER in normal clinical practice since it received marketing authorisation (27 March 2013) by the EMA OR via the compassionate use programme prior to marketing authorization.
* Where required, evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patients prescribed bosutinib as part of an interventional clinical trial programme.
* Patients initiated on bosutinib less than 3 months prior to data collection taking place.
* Patients prescribed bosutinib as exclusively post-allograft therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CML patients in a single center in Scotland.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Cumulative response rate in partial and complete haematological response (PHR/CHR) | 16 May 2019 through 30 Nov 2019
Cumulative response rate for partial and complete cytogenetic outcomes (PCyR/CCyR) | 16 May 2019 through 30 Nov 2019
Cumulative response rate for molecular response (MR) outcome | 16 May 2019 through 30 Nov 2019

SECONDARY OUTCOMES:
Proportion of patients with Philadelphia chromosome positive (Ph+) CML in chronic phase (CP), accelerated phase (AP) or blast crisis (BC) presenting with adverse events (AEs) considered related to bosutinib | 16 May 2019 through 30 Nov 2019
  AEs related to Bosutinib defined by investigator and by will be described overall (all grades of severity combined, all types of events combined) and according to grade (1,2,3 and 4 and grade 3 / 4) and by type of event
Progression-free survival | From initiation of bosutinib to 1 year, 2 year, and 3 year
  Progression will be defined as change from chronic to accelerated phase or to blast crisis.
Overall survival | From initiation of bosutinib treatment to date of death up to 30 Nov 2019
  Overall survival will be defined as the duration between initiation of bosutinib and date of death (all causes combined) (Kaplan Meier method)
The proportion of patients converting to AP/BC | 16 May 2019 through 30 Nov 2019
Proportion of patients who permanently discontinued treatment with bosutinib following an AE considered as related to bosutinib | 16 May 2019 through 30 Nov 2019
Rate of cross-intolerance between bosutinib and previously prescribed tyrosine kinase inhibitors (TKIs) | 16 May 2019 through 30 Nov 2019
  Cross-intolerance will be defined as the number of patients who permanently discontinued bosutinib because of an AE which resulted in discontinuation of a previous treatment (imatinib, dasatinib, nilotinib).
  Cross-intolerance will be estimated for all AEs, but also by type of AEs.
Mean dosage prescribed at time of initiation and mean dosage during treatment | 16 May 2019 through 30 Nov 2019
Proportion of patients with an increase or reduction in dose | 16 May 2019 through 30 Nov 2019
Mean and relative dose intensity | 16 May 2019 through 30 Nov 2019
  Defined as result of ratio of dose received over expected dose.
Proportion of patients who temporarily discontinued treatment | 16 May 2019 through 30 Nov 2019
Proportion of patients who permanently discontinued | 16 May 2019 through 30 Nov 2019
Duration of treatment | 16 May 2019 through 30 Nov 2019
  Duration of initiation up to end of treatment will be calculated for all causes of discontinuation combined and according to cause for discontinuation.
Describe the reason for selection of bosutinib in second line CML setting | 16 May 2019 through November 2019
  Clinician reason given for selecting Bosutinib therapy

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- eatson West of Scotland Cancer Centre, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1871058